CLINICAL TRIAL: NCT01479647
Title: A Phase 1, Randomized, Open-Label, Single Dose, 2-Cohort Crossover Study To Determine The Effect Of Food On The Pharmacokinetics Of Orally Administered PH-797804 In Healthy Volunteers
Brief Title: A Study To Investigate The Effect Of Food On The Pharmacokinetics Of PH-797804
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6631034
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PH 797804

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- PH-797804 1 mg Fasted (Experimental): Subjects will receive a single 1 mg dose in the fasted state
  Interventions: Drug: PH-797804
- PH-797804 1 mg Fed (Experimental): Subjects will receive a single 1 mg dose following a high-fat meal
  Interventions: Drug: PH-797804
- PH-797804 10 mg Fasted (Experimental): Subjects will receive a single 10 mg dose in the fasted state
  Interventions: Drug: PH-797804
- PH-797804 10 mg Fed (Experimental): Subjects will receive a single 10 mg dose following a high-fat meal
  Interventions: Drug: PH-797804
- PH-797804 24 mg Fed (Experimental): Subjects will receive a single 24 mg dose following a high-fat meal
  Interventions: Drug: PH-797804

INTERVENTIONS:
Drug: PH-797804 — Tablet, 1 mg, single dose
  Arms: PH-797804 1 mg Fasted
Drug: PH-797804 — Tablet, 1 mg, single dose
  Arms: PH-797804 1 mg Fed
Drug: PH-797804 — Tablet, 10 mg, single dose
  Arms: PH-797804 10 mg Fasted
Drug: PH-797804 — Tablet, 10 mg, single dose
  Arms: PH-797804 10 mg Fed
Drug: PH-797804 — Tablet, 24 mg, single dose
  Arms: PH-797804 24 mg Fed

SUMMARY:
The purpose of this study is to investigate the effect of food on the time course of PH-797804 concentration in the blood following dosing by oral immediate release tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects of non-child bearing potential between the ages of 21 and 55 years (inclusive). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: peak plasma concentration | 0,1,2,3,4,6,8,12,24,48,72,96,144,192,264,312 hours post-dose
Pharmacokinetics: time to peak plasma concentration | 0,1,2,3,4,6,8,12,24,48,72,96,144,192,264,312 hours post-dose
Pharmacokinetics: area under the plasma concentration-time curve | 0,1,2,3,4,6,8,12,24,48,72,96,144,192,264,312 hours post-dose
Pharmacokinetics: terminal plasma half-life | 0,1,2,3,4,6,8,12,24,48,72,96,144,192,264,312 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631034&StudyName=A%20Study%20To%20Investigate%20The%20Effect%20Of%20Food%20On%20The%20Pharmacokinetics%20Of%20PH-797804